CLINICAL TRIAL: NCT07053969
Title: The Effect Of Enamel Matrix Derivatives On Gingival Tissue Thickness. A Randomized Controlled Trial.
Brief Title: The Effect Of Enamel Matrix Derivatives On Gingival Tissue Thickness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Angela Palaiologou-Gallis, DDS, MS, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001758
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dental Implantation; Missing Teeth; Periodontitis, Adult; Mucositis
Keywords: Enamel Matrix Derivatives; EMD; Keratinized mucosa width; Mucosal thickness
MeSH Terms: conditions — Anodontia; Chronic Periodontitis; Mucositis

STUDY DESIGN:
Intervention Model Description: A two-arm randomized controlled trial
Who Masked: Participant
Masking Description: Prior to the beginning of the surgical procedure, the PI will request that a faculty member not involved in the case randomly select a sealed envelope and hand it to the resident completing the procedure. The surgeon will not be blinded as it is not possible since only the experimental group will only receive the EMD.The patients will be blinded as to which group they are randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1: Experimental Group using EMD (Experimental): During implant uncovering the experimental group will receive EMD under the buccal flap
  Interventions: Device: Enamel Matrix Derivative
- Group 2: Control Group (No Intervention): No EMD is administered under the buccal flap during suturing

INTERVENTIONS:
Device: Enamel Matrix Derivative — EMD is an FDA approved medical device used in periodontal procedures since 1996. It has been shown to enhance soft and hard tissue healing, increased root coverage and aid in periodontal regeneration. It's use as an adjunct during implant uncovering may increase peri-implant mucosal thickness.
  Other Names: EMD
  Arms: Group 1: Experimental Group using EMD

SUMMARY:
Scientists do research to answer important questions which might help change or improve the way we do things in the future.

The investigators know that using Enamel Matrix Derivatives results in thicker gum tissues around teeth. This study will test to see if using EMD around implants results in thicker gum tissues around implants.

DETAILED DESCRIPTION:
The hypothesis of the study is that the addition of EMD under the gingival flap prior to suturing will result in increased mucosal tissue thickness and increased keratinized tissue width as compared to not using the EMD.

The EMD will be deposited under the mucosal flap during the second stage implant uncovering. After flap suturing, an intraoral scan will be obtained. This procedure will require approximately 5 - 10 minutes per patient. All patients will be followed up at 14 days for suture removal per standard of care and not as part of the study. All patients will be followed up at one and three months per standard of care during which visits they will undergo an intraoral scan to allow evaluation of soft tissue dimensions. This is research only procedure that is expected to add 5 - 10 minutes to the regular postoperative visit. Study participation will be completed at the 3-month visit.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Males and females; Age 18 to 89 years old
3. Require second stage implant uncovering
4. In either the maxillary or mandibular arch
5. Has consistent transportation for all clinical and study visits

Exclusion Criteria:

1. Pregnancy, or those planning to become pregnant
2. Allergy or any medical issue using EMD
3. Non-English speaking
4. Patients on anticoagulants
5. Patients who object to the use of animal products

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mucosal Thickness | One month and 3 months
  Mucosal thickness at 1 and 5mm below the free gingival margin will be measured
Change in Keratinized mucosal width | One month and 3 months
  measurement of keratinized mucosal width at one and three months after surgical uncovering of the dental implant

CONTACTS AND LOCATIONS:
Overall Officials: Angela Palaiologou-Gallis, DDS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented as appropriate.
Supporting Information: Study Protocol, SAP
Time Frame: At the conclusion of the study after data analysis is complete and the research is published in a peer reviewed journal